CLINICAL TRIAL: NCT03690323
Title: Pancreatic Locally Advanced Irresectable Cancer Ablation; a Randomized Controlled Superiority Phase III Multicenter Trial
Brief Title: Pancreatic Locally Advanced Irresectable Cancer Ablation
Acronym: PELICAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Dutch Cancer Society (Other); Comprehensive Cancer Centre The Netherlands (Other); Olympus (Industry)
Responsible Party: Principal Investigator, I.Q. Molenaar, Professor, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL50467.018.14
Record Dates: First submitted 2018-09-25; First posted 2018-10-01 (Actual); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: Locally Advanced Pancreatic Cancer
Keywords: Pancreatic cancer; Pancreatic neoplasms; Locally advanced pancreatic cancer; Radiofrequency ablation; Chemotherapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiofrequency Ablation; folfirinox; 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Intervention Model Description: Radiofrequency ablation (RFA) plus chemotherapy versus chemotherapy monotherapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RFA (Experimental): RFA: laparotomy is performed followed by radiofrequency ablation of the tumor.
  After recovery of the RFA patients will continue chemotherapy:
  FOLFIRINOX or nab-paclitaxel + gemcitabine or gemcitabine monotherapy
  Interventions: Procedure: Radiofrequency ablation (RFA); Drug: FOLFIRINOX; Drug: Nab-paclitaxel plus Gemcitabine; Drug: Gemcitabine
- Chemotherapy (Active Comparator): Patients will continue chemotherapy:
  FOLFIRINOX or nab-paclitaxel plus gemcitabine or gemcitabine monotherapy
  Interventions: Drug: FOLFIRINOX; Drug: Nab-paclitaxel plus Gemcitabine; Drug: Gemcitabine

INTERVENTIONS:
Procedure: Radiofrequency ablation (RFA) — RFA involves the implantation of electrodes directly into the tumor, with the use of intra-operative ultrasound. The electrodes produce a high frequency alternating current, which leads to frictional heating and thus tissue destruction by thermal coagulation and protein denaturation.
  Other Names: Celon ProSurge bipolar probe
  Arms: RFA
Drug: FOLFIRINOX — Oxaliplatin 85mg/m2 given as 2-hour IV infusion, followed by leucovorin 400mg/m2 given as 2-hour IV infusion with addition of irinotecan 180mg/m2 given as 90-minute IV infusion. Followed by fluorouracil 400mg/m2 IV bolus, followed by continuous IV infusion of 2400mg/m2 during 46-hour. Every 2 weeks.
Drug: Nab-paclitaxel plus Gemcitabine — Nab-paclitaxel 125mg/m2 given as 30-40-minute IV infusion, followed by gemcitabine 1000mg/m2 IV infusion. On day 1, 8 and 15 every 4 weeks.
Drug: Gemcitabine — Gemcitabine 1000mg/m2 given as 30-minute IV infusion. On day 1, 8 and 15 every 4 weeks.

SUMMARY:
The aim of the PELICAN trial is to investigate the survival benefit of RFA plus standard palliative chemotherapy as compared to palliative chemotherapy alone in patients with LAPC after 2 months of induction chemotherapy.

DETAILED DESCRIPTION:
Pancreatic cancer is the fifth leading cause of cancer-related death in the Netherlands. Each year around 900 patients in the Netherlands are diagnosed with irresectable locally advanced pancreatic cancer (LAPC), which has a median survival of 7.9 months. Standard treatment is palliative chemotherapy, which offers only a very limited survival benefit. Radiofrequency ablation (RFA) is a new ablative technique for LAPC, which is feasible and safe and has been suggested to improve survival. A randomized controlled trial has not yet been performed.

The aim of the PELICAN trial is to investigate the survival benefit of RFA plus standard palliative chemotherapy as compared to palliative chemotherapy alone in patients with LAPC after 2 months of induction chemotherapy. In a randomized controlled parallel-group superiority multicenter phase III clinical trial.

The intervention will be RFA followed by chemotherapy (gemcitabine monotherapy, nab-paclitaxel plus gemcitabine or FOLFIRINOX). The comparison will be standard palliative treatment consisting of gemcitabine monotherapy, nab-gemcitabine plus gemcitabine or FOLFIRINOX Primary endpoint: Overall survival. Secondary endpoints: Progression free survival, complications, pain, radiological tumor response, CA-19.9 and CEA response, quality of life, immunomodulation and total direct and indirect costs.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed adenocarcinoma of the pancreas
2. Locally irresectable tumor
3. Primary tumor
4. Stable disease or partial response after 2 months of induction chemotherapy (according to RECIST)
5. Fit for chemotherapy as assessed by the medical oncologist, plus:

   * Absolute neutrophil count: 1.5 × 109/L
   * Platelet count: 100 × 109/L
   * Renal function: creatinine clearance> 50 ml/min
   * Transaminases ≤ 3 x ULN
6. Fit for surgery assessed by the treating surgeon and anesthesiologist
7. RFA technical feasible
8. Written informed consent
9. Age ≥ 18 years
10. Expert panel approval for randomisation

Exclusion Criteria:

1. WHO performance status ≥ 3
2. Distant metastases on abdominal or thoracic CT scan*
3. Previous surgical, local ablative or radiotherapy for pancreatic cancer or chemotherapy which is inconsistent with the prescribed induction schedule according to protocol**
4. Stenosis of > 50% of the hepatic artery AND stenosis of >50% of the portal vein/ superior mesenteric vein
5. Second primary malignancy, except adequately treated non-melanoma skin cancer, in situ carcinoma of the cervix uteri or other malignancies treated at least 5 years previously without signs of recurrence.
6. Pregnancy

   * Positive regional lymph nodes metastases are not a reason for exclusion. Lymph nodes are considered as regional, according to the consensus statement by the International Study Group of Pancreatic Surgery (ISGPS). Suspicious lymph nodes only on radiologic basis are not considered as metastasis. Only when suspicion is high due to large infiltration, pathological examination by FNA can be considered.

     * Surgical exploration is not a contra-indication for inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Estimated)
Dates: Start 2015-04-07 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 1.5 years
  The period of time between randomization and death from any cause

SECONDARY OUTCOMES:
Progression free survival | 1.5 years
  The period of time between randomization and disease progression or death (by any cause)
Complications | 1.5 years
  The occurence of any post-operative complications
Radiological tumor response | 1.5 years
  The radiologic tumor response between start of study treatment till end of follow up (or death)
Tumor marker response | 1.5 years
  The response of the tumor marker between start of study treatment till end of follow up (or death)
Quality of Life questionnaire | 1.5 years
  The quality of life measured between start study treatment till end of follow up (or death)

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Amsterdam UMC, Amsterdam, North Holland
  - Regionaal Academisch Kankercentrum Utrecht, Utrecht

REFERENCES:
- [Derived] Walma MS, Rombouts SJ, Brada LJH, Borel Rinkes IH, Bosscha K, Bruijnen RC, Busch OR, Creemers GJ, Daams F, van Dam RM, van Delden OM, Festen S, Ghorbani P, de Groot DJ, de Groot JWB, Haj Mohammad N, van Hillegersberg R, de Hingh IH, D'Hondt M, Kerver ED, van Leeuwen MS, Liem MS, van Lienden KP, Los M, de Meijer VE, Meijerink MR, Mekenkamp LJ, Nio CY, Oulad Abdennabi I, Pando E, Patijn GA, Polee MB, Pruijt JF, Roeyen G, Ropela JA, Stommel MWJ, de Vos-Geelen J, de Vries JJ, van der Waal EM, Wessels FJ, Wilmink JW, van Santvoort HC, Besselink MG, Molenaar IQ; Dutch Pancreatic Cancer Group. Radiofrequency ablation and chemotherapy versus chemotherapy alone for locally advanced pancreatic cancer (PELICAN): study protocol for a randomized controlled trial. Trials. 2021 Apr 29;22(1):313. doi: 10.1186/s13063-021-05248-y. PMID 33926539